CLINICAL TRIAL: NCT04325581
Title: Effect of Laparoscopic Sleeve Gastrectomy and Liraglutide on Glucose Homeostasis and Intrapancreatic Fat in Obese Patients
Brief Title: Laparocopic Sleeve Gastrectomy With or Without Liraglutide in Obese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: pgi123
Record Dates: First submitted 2020-03-20; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Liraglutide; Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Interventional , Placebo Control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post LSG with Liraglutude (Experimental): Liraglutide in incremental dose upto maximum of 1.8 mg per day subcutaneously once a day.
  Interventions: Drug: Liraglutide 6 MG/ML
- Post LSG without Liraglutide (Placebo Comparator): Normal Saline in equivalent per day subcutaneously once a day
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Liraglutide 6 MG/ML — Liraglutide in incremental dose upto maximum of 1.8 mg per day SC daily
  Other Names: Calorie restricted diet
  Arms: Post LSG with Liraglutude
Drug: Placebos — Normal Saline SC daily
  Other Names: Calorie restricted diet
  Arms: Post LSG without Liraglutide

SUMMARY:
Investigators postulate that the metabolic effects of LSG would be augmented with the use of liraglutide leading to additional excess weight loss, improved glucose homeostasis, decreased intrapancreatic and intrahepatic fat than either of them individually. However there are no studies till date which have evaluated the combined effects of two modalities of weight loss on the above mentioned parameters. This study plans to compare the effects of liraglutide in post- LSG obese patients in a placebo controlled design.

DETAILED DESCRIPTION:
Various studies have shown that bariatric surgery is associated with significant durable weight loss with associated improvement in obesity related comorbidities and quality of life. The degree of effect on obesity related comorbidities depends on the bariatric surgery approach, typically classified as restrictive and/or malabsorptive effect. Data from International Federation for the Surgery of Obesity and Metabolic Diseases states that most common surgical procedures being performed are Roux-en-Y gastric bypass (45%), sleeve gastrectomy(37%), adjustable gastric banding(10%) and biliopancreatic division with or without duodenal switch(2.5%)5. . LSG is technically a simpler procedure compared to RYGB with lesser operative and long term nutritional complications. The mechanism for weight loss in laparoscopic sleeve gastrectomy is gastric restriction and possible changes in gut hormones resulting from higher level of GLP-1, and lower levels of ghrelin, as a consequence of resection of gastric fundus.

Therefore,investigators postulate that the metabolic effects of LSG would be augmented with the use of liraglutide leading to additional excess weight loss, improved glucose homeostasis, decreased intrapancreatic and intrahepatic fat than either of them individually. However there are no studies till date which have evaluated the combined effects of two modalities of weight loss on the above mentioned parameters. This study plans to compare the effects of liraglutide in post- LSG obese participants in a placebo controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with obesity who have elected to undergo bariatric surgery
* Body mass index greater than 27.5kg/mt2
* Ability and willingness to co-operate with follow up.

Exclusion Criteria:

Decompensated liver disease ( child-turcotte pugh score >7)

* Impaired renal function, defined as eGFR< 45 ml/min/m2
* Clinically significant active cardiovascular disease including history of myocardial infarction within the past 6 months and/or heart failure (New York Heart Association (NYHA) class III and IV)
* Recurrent major hypoglycemic episodes
* Use of drugs like systemic corticosteroids, thiazolidinediones, DPPIV inhibitors
* Pregnancy or lactation
* History of pancreatitis or pancreatic cancer
* History of medullary thyroid cancer
* Family history of medullary thyroid cancer
* Contraindications to liraglutide or any of its excipients
* Hypersensitivity to liraglutide or similar drugs
* Patients currently using GLP-1 analogs
* Suspected or known abuse of alcohol
* Presence of secondary cause of obesity.
* Presence of an eating disorder or other psychiatric disorder.
* Prior gastric surgery.
* Unfit for surgery due to severe cardiac, pulmonary diseases or due to any reason.
* Contraindications to MRI scanning

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incretin change | baseline and at 6weeks and 6months after laparoscopic sleeve gastrectomy
  Changes in GLP-1 levels during 2hour OGTT
Changes in indices of insulin resistance | baseline and at 6weeks and 6months after laparoscopic sleeve gastrectomy
  HOMA-IR calculated from fasting insulin and fasting glucose
Change in pancreatic steatosis | baseline and 6months after laparoscopic sleeve gastrectomy
  Change in pancreatic steatosis would be determined using NUTS ACORN NMR software

SECONDARY OUTCOMES:
body weight | baseline and 6 weeks, 12weeks, 18weeks and 24weeks after surgery
  The change in body weight